CLINICAL TRIAL: NCT05367466
Title: Evaluation of Acquired and Hereditary Risk Factors of Neonatal Thrombosis: Single-centre Experience
Brief Title: Risk Factors of Neonatal Thrombosis
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Nilufer Guzoglu, Assoc. Prof, Kırıkkale University
Other Study IDs: 2022.03.38
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Thrombosis
Keywords: newborn, hereditary risk factors
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborn with thrombossis: All admitted newborns in NICU during the study period

SUMMARY:
The incidence of symptomatic thrombosis is between 2.4 and 6.8 per 1000 neonatal intensive care unit admission while it is 5.1 per 100 000 live births. Compared to adults, the anticoagulant and fibrinolytic system of newborns is significantly different.

In this study, the aim is to evaluate infants with neonatal thrombosis in our unit to characterize acquired and genetic risk factors, the laboratory work-up parameters and the diagnosis approach.

DETAILED DESCRIPTION:
All newborn patients diagnosed with neonatal thrombosis in our NICU between 2014 and 2019; were included in the study.

Patients' data: maternal and neonatal characteristics, consanguinity, need for resuscitation, Apgar scores, diagnoses, need for mechanical ventilation, sepsis, catheter placement, treatment regimens and hospital outcomes; Laboratory findings: CBC; D-dimer levels and the performed genetic test Thrombosis diagnosis was confirmed by imaging techniques such as ultrasonography (USG), echocardiography, and magnetic resonance imaging (MRI).

The genotypes: Factor V (Leiden) G1691A, prothrombin G20210A, MTHFRC677T, MTHFRA1298C, PAI-SERPINE1, Factor XIII V34L mutations

ELIGIBILITY:
Inclusion Criteria:

* All newborn accepted at NICU

Exclusion Criteria:

* No

Min Age: 1 Day | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All newborns in NICU during 5 year period
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Thrombosis in the neonatal period is multifactorial | January 2022
Hereditary thrombophilia factors also should be thought | January 2022

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guzoglu N, Albayrak M, Aliefendioglu D. Evaluation of Patients with Neonatal Thrombosis. Indian J Pediatr. 2023 Jun;90(6):615-617. doi: 10.1007/s12098-023-04497-w. Epub 2023 Mar 2. PMID 36859514